CLINICAL TRIAL: NCT04280393
Title: Effectiveness And Safety Of The Colonoscopy Assisted By Endocuff Visio Vs. Standard Colonoscopy In The Colorectal Cancer Screening Program: Clinical Random, Prospective, Multicentric, Open And Parallel Groups
Brief Title: Effectiveness and Safety of the Colonoscopy Assisted by Endocuff vs. Standard in the Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Provincial de Castellon (Other)
Responsible Party: Principal Investigator, Fernando Sabado Marti, Principal Investigator, Hospital Provincial de Castellon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: FCVHPC-2018-PS-01
Record Dates: First submitted 2020-02-14; First posted 2020-02-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Cancer Colorectal
Keywords: adenoma; colonoscopy; endocuff; screening
MeSH Terms: conditions — Colonic Neoplasms; Adenoma | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endocuff (Experimental): Colonoscopy procedure with the use of endocuff
  Interventions: Device: Colonoscopy procedure with endocuff
- Control (Active Comparator): Standard Colonoscopy procedure
  Interventions: Device: Colonoscopy procedure with endocuff

INTERVENTIONS:
Device: Colonoscopy procedure with endocuff — Colonoscopy procedure with the use of ENDOCUFF VISION

SUMMARY:
The hypothesis of the present study is to demonstrate that ENDOCUFF VISION® increases the detection rate of adenomas thanks to the improved visibility produced by the retraction of the folds and stabilizing the colonoscope. Likewise, the impact of the use of ENDOCUFF VISION® on the average number of adenomas detected per patient (MAPP) as well as serrated adenomas (MASPP), the total time of the endoscopic procedure, cecal intubation and the safety of its use will be estimated.

DETAILED DESCRIPTION:
The main objective of the colorectal cancer screening program (CRC) is the detection of the greatest number of precursor lesions of neoplasms as well as cancerous lesions established in the general population with an intermediate risk of presenting CRC. Within this program, colonoscopy is considered the diagnostic technique of choice due to its cost-effectiveness balance. However, it remains a technique that is not entirely perfect since the omission of injuries during the procedure constitutes the main reason for the appearance of interval cancers, with a clear correlation between the rate of detection of adenomas and their appearance.

The vast majority of CRC arise from precancerous polyps, of which there are two main types: conventional adenomas and serrated polyps. Conventional adenomas are the most frequent polyps being responsible for the majority of CRC through the adenoma-carcinoma sequence. It should be taken into account that about 15-30% of sporadic CRC develops from serrated polyps through the serrated pathway of carcinogenesis, which is different from the traditional adenoma-carcinoma sequence. Endoscopic detection of serrated polyps is difficult due to their indistinguishable edges and flat or sessile morphology. In addition, they tend to be located in the right colon, a place that can be more difficult to reach in colonoscopy and examine completely.

Therefore, the ultimate goal of CRC screening colonoscopy is to reduce the appearance of CRC, trying to maximize the detection of polyps and therefore the detection rate of adenomas. For this there are several technical factors of colonoscopy, preparation, imaging and external devices that try to achieve an increase in the rate of detection of adenomas.

ENDOCUFF VISION® (Norgine Pharmaceuticals Ltd) is a medical device that is fixed at the distal end of the endoscope, improving its insertion in the intestine thanks to the action it exerts by flattening the folds and stabilizing the device. Its use is related to greater accuracy in the detection of adenomas, since it increases the visibility of the mucosa and thus decreases the number of polyps that may go unnoticed, increasing the detection rate of adenomas between 10 and 16 percentage points, according with published literature .

Thus, the hypothesis of the present study is to demonstrate that ENDOCUFF VISION® increases the detection rate of adenomas thanks to the improved visibility produced by the retraction of the folds and stabilizing the colonoscope. Likewise, the impact of the use of ENDOCUFF VISION® on the average number of adenomas detected per patient (MAPP) as well as serrated adenomas (MASPP), the total time of the endoscopic procedure, cecal intubation and the safety of its use will be estimated.

ELIGIBILITY:
Inclusion Criteria:

A) Patients between the ages of 50 and 70 referred for a colonoscopy within the colorectal cancer screening program.

B) With the ability to provide informed consent

Exclusion Criteria:

1. History of inflammatory bowel disease
2. History or suspected obstruction or intestinal pseudo-obstruction located in the colon
3. History of colon cancer or polyposic syndromes
4. History of colonic stenosis
5. History of severe diverticular segments in some region of the colon
6. Subjects unable to provide informed consent
7. Subjects under treatment with clopidogrel, warfarin, acenocoumarol or other new generation anticoagulants that have not discontinued treatment in accordance with the provisions of these procedures
8. Pregnants females
9. Subjects who are going to undergo a therapeutic or surveillance endoscopy for follow-up of injuries diagnosed in previous procedures
10. Subjects whose baseline status does not allow the completion of the questionnaires necessary for the evaluation of the study objectives.
11. History of previous colonic surgery except for appendectomy
12. Any medical, psychological, psychiatric, geographic or social problem that is important and uncontrolled that may interfere with the patient's participation in the study or that does not allow adequate follow-up and adherence to the protocol and evaluation of the study results.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 822 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
polyps detection rate per patient | immediately after the procedure
  Rate of polyps detected
adenoma detection rate per patient | immediately after the procedure
  Rate of Adenoma detected

SECONDARY OUTCOMES:
differences in the mean of adenomas detected by patient | immediately after the procedure
  Assess whether there are differences in the mean of adenomas detected by patient comparing Endocuff Colonoscopy and Standard Colonoscopy.
Serrated adenoma rate detected by patient | immediately after the procedure
  Rate of serrated adenomas
Cancer lesion detection rate comparing Endocuff Colonoscopy and Standard Colonoscopy. | immediately after the procedure
  Rate of lessions
Cecal intubation rate and time to reach the cecum | immediately after the procedure
  Time in minutes of the intubation
Total time of the procedure | immediately after the procedure
  Total time of the procedure, from the insertion of the colonoscope to its extraction comparing Endocuff Colonoscopy and Standard Colonoscopy.
Colonoscope withdrawal time from cecum | immediately after the procedure
  Colonoscope withdrawal time from cecum in patients in whom no polyps were detected
Demonstrate the non-inferiority of patient experience when comparing Endocuff Colonoscopy and Standard Colonoscopy | through study completion, an average of 3 months
  Number of Participants With Procedure-Related Adverse Events Intra and post-procedure (evaluated with CTC AE v4) comparing Endocuff Colonoscopy and Standard Colonoscopy. This will be calculated as a Rate of Intra and post-procedure complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Provincial de Castellon, Castellon, Castellon, Spain

IPD SHARING:
Plan to Share IPD: No